CLINICAL TRIAL: NCT03563937
Title: Real-world Comparative Effectiveness of Stroke Prevention in Patients With Atrial Fibrillation Treated With Factor Xa Non-vitamin-K Oral Anticoagulants (NOACs) vs. Phenprocoumon
Acronym: ReLoaDeD
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 20031
Record Dates: First submitted 2018-06-11; First posted 2018-06-20 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Phenprocoumon; apixaban; Rivaroxaban; edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Phenprocoumon: Patients with NVAF who initiated the treatment of Phenprocoumon.
  Interventions: Drug: Phenprocoumon
- Apixaban: Patients with NVAF who initiated the treatment of Apixaban.
  Interventions: Drug: Apixaban
- Rivaroxaban (Xarelto, BAY59-7939): Patients with NVAF who initiated the treatment of Rivaroxaban.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Edoxaban: Patients with NVAF who initiated the treatment of Edoxaban.
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Phenprocoumon — Follow the physician's prescription.
  Groups: Phenprocoumon
Drug: Apixaban — 2.5 mg or 5 mg, twice daily
  Groups: Apixaban
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 15 mg or 20 mg, once daily
  Groups: Rivaroxaban (Xarelto, BAY59-7939)
Drug: Edoxaban — 30 mg or 60 mg, once daily
  Groups: Edoxaban

SUMMARY:
Existing real-world studies have provided evidence that novel oral anticoagulants (NOACs) in general and rivaroxaban in particular are more effective and at least as safe as warfarin in non-valvular atrial fibrillation (NVAF) patients with renal impairment. Nevertheless, it is known that clinicians often hesitate to prescribe NOACs to patients with even moderate renal impairment. Therefore, it is important to investigate effectiveness and safety of rivaroxaban and other NOACs compared to vitamin-K antagonists in NVAF patients with renal dysfunction in real life setting.

The primary objectives of this study are to describe the risk of ischemic stroke (IS)/ systemic embolism (SE) and intracranial hemorrhage (ICH) in patients with non-valvular atrial fibrillation (NVAF) and renal impairment initiating treatment with individual NOACs (rivaroxaban, apixaban, edoxaban) compared to phenprocoumon.

ELIGIBILITY:
Inclusion Criteria:

* First NOAC (rivaroxaban, apixaban, edoxaban) or phenprocoumon prescription (index drug) in the enrollment period between 1st January 2013 to 30th June 2017 (index date).
* Age of at least 18 years at index date.
* Continuous enrollment in the 12 months before the first NOAC (rivaroxaban, apixaban, edoxaban) or phenprocoumon prescription in the enrollment period (baseline period).
* A verified ambulatory or primary/ secondary hospital discharge diagnosis of NVAF in the 12 months before the first NOAC (rivaroxaban, apixaban, edoxaban) or phenprocoumon prescription in the enrollment period (baseline period).

Exclusion Criteria:

* A verified ambulatory or primary/ secondary hospital discharge diagnosis of valvular atrial fibrillation, indicating pregnancy, transient cause of atrial fibrillation or venous thromboembolism (VTE).
* A claim for hip or knee replacement surgery in the 60 days prior to or on the index date.
* A prescription of more than one oral anticoagulant (rivaroxaban, apixaban, edoxaban or phenprocoumon) on the index date.
* A prescription of warfarin or dabigatran in the baseline period or on the index date.
* A verified ambulatory or primary/ secondary hospital discharge diagnosis of end-stage kidney disease or a claim for dialysis in the baseline period.
* Patients receiving an initial dose of rivaroxaban 10 mg/ 2.5 mg or edoxaban 15 mg (these dosages are not indicated for the treatment of NVAF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population of this study will include all insured members of approximately 64 German statutory health insurances (SHIs) contributing data to the InGef database.
Sampling Method: Non-Probability Sample
Enrollment: 64920 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Risk of Ischemic stroke (IS) / Systemic embolism(SE) (as combined endpoint and alone), recurrent IS/SE (as combined endpoint) and severe IS in patients with NVAF and renal impairment determined by inpatient claims based diagnoses | Retrospective analysis from January 2012 - December 2017
  Severe IS will be defined according to an approach proposed by Schubert et al. as hospitalization with a primary hospital discharge diagnosis of IS in combination with an OPS (Operationen und Prozedurenschlüssel) code indicating one of the following: intubation, mechanical ventilation or percutaneous endoscopic gastronomy
Risk of intracranial hemorrhage (ICH) in patients with non-valvular atrial fibrillation (NVAF) with renal impairment determined by inpatient claims based diagnoses | Retrospective analysis from January 2012 - December 2017
Healthcare resource consumption in patients with non-valvular atrial fibrillation (NVAF) and renal impairment determined by inpatient claims based diagnoses | Retrospective analysis from January 2012 - December 2017
Overall costs in patients with renal impairment determined by inpatient claims based diagnoses | Retrospective analysis from January 2012 - December 2017
Sector specific costs in patients with renal impairment determined by inpatient claims based diagnoses | Retrospective analysis from January 2012 - December 2017

SECONDARY OUTCOMES:
Risk of fatal bleeding in patients with NVAF (overall population as well as patients with renal impairment) determined by inpatient claims based diagnoses | Retrospective analysis from January 2012 - December 2017
  Fatal bleeding will be defined as hospitalization with a primary hospital discharge diagnoses for bleeding with documented death as reason for hospital discharge or within 30 days after hospital discharge.
Risk of recurrent hospitalizations (in general and for IS/SE) | Retrospective analysis from January 2012 - December 2017
Risk of Kidney failure determined by inpatient claims based diagnoses | Retrospective analysis from January 2012 - December 2017
Risk of Acute kidney injury (AKI) determined by inpatient claims based diagnoses | Retrospective analysis from January 2012 - December 2017
Risk of treatment discontinuation in patients with NVAF (overall population as well as patients with renal impairment) determined by pharmacy claims | Retrospective analysis from January 2012 - December 2017
Risk of IS, SE, Severe IS and recurrent IS/SE in patient with NVAF determined determined by inpatient claims based diagnoses | Retrospective analysis from January 2012 - December 2017

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Germany